CLINICAL TRIAL: NCT06998420
Title: Construction of a Clinical Prediction Model for Poor Prognosis Following Percutaneous Balloon Compression of the Trigeminal Ganglion
Brief Title: Developing a Clinical Prediction Model for Adverse Outcomes in Percutaneous Trigeminal Ganglion Balloon Compression
Status: Completed | Type: Observational
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-K098-01
Record Dates: First submitted 2025-05-08; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-02

CONDITIONS: Trigeminal Neuralgia (TN)
Keywords: Trigeminal neuralgia; PCGG; poor prognosis; Clinical Prediction Model
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This clinical study aims to investigate adverse outcomes following percutaneous balloon compression (PBC) of the trigeminal ganglion, establish a predictive model, and assess the probability of postoperative complications.The main question it aims to answer is:

1. What factors are associated with adverse postoperative outcomes?
2. What is the occurrence probability of different types of adverse outcomes? The study will record patients' demographic and clinical characteristics, laboratory test results, and conduct follow-ups at 3, 6, and 12 months postoperatively.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosed with primary trigeminal neuralgia and underwent PBCG at the Pain Department of Affiliated Hospital of Nantong University
2. Age ≥18 years
3. Willing to complete postoperative follow-up

Exclusion criteria:

1. Secondary trigeminal neuralgia (e.g., tumor compression, multiple sclerosis)
2. Previous interventional treatments for trigeminal neuralgia
3. Incomplete follow-up data
4. General anesthesia contraindications or significant dysfunction of major organs (cardiac, pulmonary, hepatic, renal) or severe neurological impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent PCGG surgery at the Pain Department of Affiliated Hospital of Nantong University between 2022 and 2024 and were willing to participate in postoperative follow-up were selected as the study subjects.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Pain recurrence (BNI≥Ⅲ) | Follow-up timepoints: 3, 6, and 12 months postoperatively (final determination based on preliminary observation endpoints)
  BNI Pain Intensity Scale Score:
  I:No pain,no medication II:Occasional pain,not requiring medication III:Some pain,adequately controlled with medication IV:Some pain,not adequately controlled with medication V:Severe pain/no pain relief
Severe sensory impairment (facial numbness with BNI sensory score ≥ Grade III) | 3 months, 6 months, and 12 months postoperatively (determined based on prior observation endpoints).
  BNI Pain Intensity Scale Score:
  I:No pain,no medication II:Occasional pain,not requiring medication III:Some pain,adequately controlled with medication IV:Some pain,not adequately controlled with medication V:Severe pain/no pain relief
Masticatory dysfunction (bite force reduction ≥50% or subjective weakness) | 3 months, 6 months, and 12 months postoperatively (determined based on prior observation endpoints).

SECONDARY OUTCOMES:
Mild sensory abnormalities (BNI sensory score Grade II) | 3 months, 6 months, and 12 months postoperatively (determined based on prior observation endpoints).
  BNI Pain Intensity Scale Score:
  I:No pain,no medication II:Occasional pain,not requiring medication III:Some pain,adequately controlled with medication IV:Some pain,not adequately controlled with medication V:Severe pain/no pain relief
Diplopia or hearing loss (rare complications to be recorded) | 3 months, 6 months, and 12 months postoperatively (determined based on prior observation endpoints).
Postoperative infection (puncture site/intracranial) | 3 months, 6 months, and 12 months postoperatively (determined based on prior observation endpoints).
Psychological status (change in HADS score) | 3 months, 6 months, and 12 months postoperatively (determined based on prior observation endpoints).
  he HADS (Hospital Anxiety and Depression Scale) is a self-assessment questionnaire used to screen for anxiety (HADS-A) and depression (HADS-D) in patients, with each subscale ranging from 0 (no symptoms) to 21 (severe symptoms). A score ≥8 on either subscale suggests clinically significant symptoms.
  Key features:
  14 items (7 for anxiety, 7 for depression)
  Simple & fast (takes ~5 min)
  Designed for non-psychiatric medical settings
  Example scoring:
  0-7: Normal
  8-10: Mild
  11-14: Moderate
  15-21: Severe

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Nantong University, Nantong, Jiangsu, China